CLINICAL TRIAL: NCT02552940
Title: A PROSPECTIVE, NON-INTERVENTIONAL STUDY TO EVALUATE THE CLINICAL EFFECTIVENESS, THE CONSISTENCY OF EVALUATION SCORES, QUALITY OF LIFE, SAFETY AND TOLERABILITY OF TOCILIZUMAB SUBCUTANEOUS IN PATIENTS WITH RHEUMATOID ARTHRITIS IN DAILY CLINICAL PRACTICE
Brief Title: An Observational Study to Evaluate the Clinical Effectiveness, Quality of Life, Safety and Tolerability of Tocilizumab (TCZ) in Patients With Rheumatoid Arthritis (RA) in Daily Clinical Practice
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: nv Roche sa (Unknown)
Responsible Party: Sponsor
Other Study IDs: ML29691
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rheumatoid Arthritis participants treated with Tocilizumab SC: Participants with RA receive TCZ SC, as per routine clinical practice and are followed for approximately 6 months.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Participants with RA receive TCZ SC, as per routine clinical practice and are followed for approximately 6 months.
  Other Names: RoACTEMRA

SUMMARY:
This observational trial will evaluate the effectiveness, the consistency of evaluation scores, quality of life, safety and tolerability of TCZ administered subcutaneously (SC) in participants with RA in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants naive to TCZ or who have received TCZ SC treatment within 8 weeks prior to the enrolment visit can be included
* Participants in whom the treating physician has made the decision to commence TCZ SC in accordance with the label and reimbursement criteria

Exclusion Criteria:

* Participants who have received TCZ >8 weeks prior to the enrolment visit
* Participants who have previously received TCZ SC
* Participants who have received treatment with any investigational agent within 4 weeks before starting treatment with TCZ SC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant with a diagnosis of moderate to severe RA defined as DAS28 more than or equal to (>=) 3.7, naïve to TCZ and in whom the treating physician has made the decision to commence TCZ SC in accordance with the label and reimbursement criteria
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2015-10-31 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-10-23 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient between DAS28 - erythrocyte sedimentation rate (DAS28-ESR) and Clinical Disease Activity Index (CDAl) | Up to Week 24

SECONDARY OUTCOMES:
Correlation Coefficient Between CDAI and simplified disease activity index (SDAI) and Between SDAI and DAS28-ESR | Up to Week 24
Percentage of participants to achieve low disease activity (LDA) using DAS28 (less than or equal to [<=] 3.2), CDAl (<=10.0) and SDAI (<=11 .0) | Up to Week 24
Time to achieve low disease activity (LDA) using DAS28 (<= 3.2), CDAl (<=10.0) and SDAI (<=11 .0) | Up to week 24
Percentage of participants to achieve disease remission using DAS28-ESR (<2.6), CDAl (<=2.8) and SDAI (<=3.3) | Up to Week 24
Time to achieve disease remission using DAS28-ESR (<2.6), CDAl (<=2.8) and SDAI (<=3.3) | Up to Week 24
Percentage of participants to achieve a clinically meaningful improvement in DAS28-ESR (reduction of at least 1.2 units) | Up to Week 24
Time to achieve a clinically meaningful improvement in DAS28-ESR (reduction of at least 1.2 units) | Up to Week 24
Percentage of participants to achieve a major and minor improvement in CDAl (more than or equal to [>=]13.9 and >=6.7, respectively) and SDAI (>=17.1 and >=6.9, respectively) | Up to Week 24
Time to achieve a major and minor improvement in CDAl (>=13.9 and >=6.7, respectively) and SDAI (>=17.1 and >=6.9, respectively) | Up to Week 24
Change from baseline in total tender joint count (TJC) | Up to Week 24
Change from baseline in total swollen joint count (SJC) | Up to Week 24
Percentage of participants having TJC <=1 | Up to Week 24
Percentage of participants having SJC <=1 | Up to Week 24
Patient Global Assessment of disease activity visual analogue scale (VAS) score | Up to Week 24
Physician Global Assessment of disease activity VAS score | Up to Week 24
Percentage of participants having CRP <=1mg/dl | Up to Week 24
Health Assessment Questionnaire Disability Index (HAQ-DI) | Up to Week 24
EQ-5D-5L Health Questionnaire (EuroQoL) | Up to Week 24
Morisky Medication-Taking Adherence Scale (MMAS) | Up to Week 24
Percentage of participants using TCZ in monotherapy | At baseline
Percentage of participants using TCZ in combination with disease-modifying antirheumatic drug's (DMARD's) | At baseline
Percentage of participants presenting a high inflammation (DAS28-ESR >5.1) | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- Belgium (21):
  - ASZ Aalst, Aalst
  - AZ Sint Lucas Brugge, Assebroek
  - AZ Sint Jan, Bruges
  - CHU St Pierre (César de Paepe), Brussels
  - HIS (Etterbeek Ixelles), Brussels
  - Hospital Erasme; Neurologie, Brussels
  - AZ Sint Blasius (Dendermonde), Dendermonde
  - UZ Antwerpen, Edegem
  - Reumacentrum Genk, Genk
  - Reumaclinic, Genk
  - GHdC Site Saint-Joseph, Gilly (Charleroi)
  - AZ Groeninge, Kortrijk
  - CHU Sart-Tilman, Liège
  - Private Practice, Lokeren
  - CHU UCL Mont-Godinne, Mont-godinne
  - AZ Damiaan, Ostend
  - AZ Oudenaarde, Oudenaarde
  - AZ Alma vzw (Sijsele), Sijsele
  - AZ Sint Jozef Malle, Westmalle
  - Sint Augustinus Wilrijk, Wilrijk
  - CVBA Diagnosecentrum Voorkempen, Zoersel
- Höpital Kirchberg; Rheumatology, Luxembourg, Luxembourg